CLINICAL TRIAL: NCT01561300
Title: Efficacy of Standardized Brooke Bond Black Tea Extract on Flow-Mediated Dilation After an Acute Dose as Well as After One Week of Consumption in Healthy Adult Indian Males
Brief Title: Efficacy of Brooke Bond Black Tea Extract on Flow Mediated Dilation in Indian Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: Lotus Labs Pvt. Ltd, Bangalore, India (Unknown); Clumax Diagnostics, Bangalore, India (Unknown); Quipu S.r.l, Pisa, Italy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: FDS-BEV-0284
Record Dates: First submitted 2012-03-20; First posted 2012-03-23 (Estimated); Results first posted 2017-04-05 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-02

CONDITIONS: Healthy
Keywords: Black tea; Flow Mediated Dilation; Vascular function; India
MeSH Terms: interventions — Tea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Nutrition intervention study with a control
  Interventions: Other: Nutrition intervention study with a control
- Tea extract (Experimental): Nutrition intervention study with a black tea extract
  Interventions: Other: Nutrition intervention study with a black tea extract

INTERVENTIONS:
Other: Nutrition intervention study with a black tea extract — Tea extract: 1800 mg/day standardized Brooke Bond black tea extract equivalent to 400 mg flavonoids dissolved in 240 ml hot water.
  Products will be consumed for 8 days. On measurement days tea will be given to the subjects as a single acute dose and 2 grams of sugar will be added.
  On day 2-7 subjects will consume 3 cups or tea, each prepared with 800 mg product in 80 ml of boiling water and sugar added to subject's taste. First cup of tea will be taken as morning tea, 2nd at breakfast and 3rd in the evening. No milk will be added.
  Other Names: Black tea extract
  Arms: Tea extract
Other: Nutrition intervention study with a control — Control: 1800 mg/day of a powder that gives a flavoured beverage with a color similar to black tea dissolved in 240 ml hot water.
  Products will be consumed for 8 days. On measurement days control will be given to the subjects as a single acute dose and 2 grams of sugar will be added.
  On day 2-7 subjects will consume 3 cups of control, each prepared with 800 mg product in 80 ml of boiling water and sugar added to subject's taste. First cup of tea will be taken as morning tea, 2nd at breakfast and 3rd in the evening. No milk will be added.
  Other Names: Control
  Arms: Control

SUMMARY:
This study examines the effect of 1800 mg/day standardized Brooke Bond black tea extract, equivalent to 400 mg flavonoids, on Flow Mediated Dilation in healthy Indian males.

DETAILED DESCRIPTION:
Flow mediated dilation (FMD) is a non-invasive measurement technique performed using ultrasound equipment to measure hyperaemia induced dilation of blood vessels. Evidence from prospective studies suggests that FMD is independently inversely associated with cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Male volunteers aged between >_30 _< 50 years of age
* Body Mass Index (BMI) of >_18 and _< 25.0 kg/m2
* Systolic blood pressure >_140 and >_100 mmHg and diastolic blood pressure < 90 and > 70 mmHg
* Subjects who consume _< 2 cups of coffee per day
* Subjects who drink tea regularly (>_ 2 cups per day)
* Apparently healthy, with no reported medical condition which might affect the assessment as judged by the study physician or/and PI
* No prescribed medical treatment that may affect study parameters as judged by the Study Physician
* Subject willing to abstain from alcohol on day before and on the day of assessment
* Willing to sign the informed consent form

Exclusion Criteria:

* Smokers and/or tobacco chewers
* Those who consume regular alcohol (> 160 ml of alcohol per week)
* Reported intense sport activities > 10h/week
* Participating in any other clinical study concurrently or if participated in any study during 2 months preceding the screening visit

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-03; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anisha Pargal, Dr, Study Director — Unilever Industries Pvt. Ltd
Locations (1):
- Lotus Labs Pvt. Ltd.,, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty five subjects were invited for screening. Two subjects did not come for the screening, three subjects were not willing to participate and three subjects did not fulfil the inclusion criteria. Of the 37 subjects that fulfilled all inclusion an exclusion criteria 30 were invited to participate.
Pre-assignment Details: Thirty subjects meeting all criteria were randomised over the two arms
Groups:
- Control, Then Washout, Then Tea: Subjects first received Control for one week with Flow Mediated Dilation (FMD) measurements on day 1 and day 8. After a washout of one week (day 8-15) they received Tea for one week with FMD measurements at day 16 and day 22. All FMD measurements were done in a fasted state just before test product intake and exactly 2 hours after test product intake.
- Tea, Then Wash Out, Then Control: Subjects first received Tea for one week with with Flow Mediated Dilation (FMD) measurements on day 1 and day 8. After a washout of one week (day 8-15) they received Control for one week with FMD measurements at day 16 and day 22. All FMD measurements were done in a fasted state just before test product intake and exactly 2 hours after test product intake.
Period: Run in on Placebo
Arm/Group | Control, Then Washout, Then Tea | Tea, Then Wash Out, Then Control
Started | 15 | 15
Completed | 14 | 15
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: First Intervention
Arm/Group | Control, Then Washout, Then Tea | Tea, Then Wash Out, Then Control
Started | 14 | 15
Completed | 14 | 15
Not Completed | 0 | 0
Period: Washout on Placebo
Arm/Group | Control, Then Washout, Then Tea | Tea, Then Wash Out, Then Control
Started | 14 | 15
Completed | 14 | 15
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Control, Then Washout, Then Tea | Tea, Then Wash Out, Then Control
Started | 14 | 15
Completed | 14 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Population: All participants who were randomised
Arm/Group | Study Population
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years]
  Age | 36 [30 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 30
Region of Enrollment [Number; unit: participants]
  India | 30
Body Mass Index [Median (Full Range); unit: kg/m^2] | 23.2 [18.5 to 26.4]

OUTCOME MEASURES:

1. Primary Outcome: 'Acute-upon-chronic Effect' of Tea vs Control
Description: Change in flow mediated dilation (FMD) due to tea consumption when compared to control.
  FMD measurement included the following steps:
  * 1 minute base scan to measure the baseline diameter of artery (baseline)
  * 5 minutes of forearm occlusion at 300±30 mmHg, just below the elbow 2-5 cm from antecubital crease
  * 4 minutes FMD scan, which started immediately after release of the occlusion (reactive hyperaemia stage) FMD was calculated as maximal percentage change in diameter of the artery above the baseline value after the release of the occlusion
Time Frame: Baseline day 1 to 2 hours post consumption on day 8.
Population: Per protocol based on the full data set excluding one subject who did produce relevant data (AE) and three subjects who were removed during blind review (operator comments, hypertension and increase in body weight). Single data points were removed for 6 subjects (all single data points) based on operator comments.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of change in diameter
Groups:
- Tea Beverage: Participants when they received tea
- Control Beverage: Participants when they received control
Arm/Group | Tea Beverage | Control Beverage
Number analyzed (Participants) | 27 | 27
percentage of change in diameter | 8.03 [6.95 to 9.12] | 9.03 [8.01 to 10.05]
Statistical Analysis 1: Comparison: Tea Beverage vs Control Beverage; Null hypothesis: no difference between Tea and Control; Test type: Superiority or Other; p = 0.09, Mixed Models Analysis; Subject as random factor, baseline same period and mean baseline in both periods as covariates, and treatment, operator, and period as fixed effects; Mean Difference (Final Values) = -1.00, 95% CI 2-sided [-2.16 to 0.17] — Tea-placebo

2. Secondary Outcome: Acute Effect of Tea vs Control
Description: Change in flow mediated dilation due to tea consumption when compared to control.
  FMD measurement included the following steps:
  * 1 minute base scan to measure the baseline diameter of artery (baseline)
  * 5 minutes of forearm occlusion at 300±30 mmHg, just below the elbow 2-5 cm from antecubital crease
  * 4 minutes FMD scan, which started immediately after release of the occlusion (reactive hyperaemia stage) FMD was calculated as maximal percentage change in diameter of the artery above the baseline value after the release of the occlusion
Time Frame: From baseline on day 1 to 2 hours post consumption on day 1
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change in flow mediated dilation
Arm/Group | Tea Beverage | Control Beverage
Number analyzed (Participants) | 27 | 27
percent change in flow mediated dilation | 8.44 [7.08 to 9.79] | 8.82 [7.52 to 10.09]
Statistical Analysis 1: Comparison: Tea Beverage vs Control Beverage; Null hypothesis: no difference between Tea and Control; Test type: Superiority or Other; p = 0.70, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-2.44 to 1.66] — Tea- Control

3. Secondary Outcome: Chronic Effect of Tea vs Control
Description: as for outcome 1
Time Frame: From baseline at day 1 to baseline on day 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change in flow mediated dilat
Arm/Group | Tea Beverage | Control Beverage
Number analyzed (Participants) | 27 | 27
Percentage change in flow mediated dilat | 9.19 [8.28 to 10.09] | 9.39 [8.51 to 10.27]
Statistical Analysis 1: Comparison: Tea Beverage; Null hypothesis: no difference between Tea and Control; Test type: Superiority or Other; p = 0.66, Mixed Models Analysis — Subject as random factor, baseline same period and mean baseline in both periods as covariates, and treatment, operator, and period as fixed effects; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-1.15 to 0.75] — Tea-placebo

ADVERSE EVENTS:
Groups:
- Tea Extract: Subjects when they consumed tea extract for one week
- Control: Subjects when they consumed control for one week
- Placebo: Subjects when they consumed placebo for 6 days during the run in and during 7 days during the washout
Arm/Group | Tea Extract | Control | Placebo
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 1/29 | 1/29 | 3/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tea Extract (N=29) | Control (N=29) | Placebo (N=30)
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Subject developed hypertension after being included
Upper restiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) — During tea drinking
Increased ferquency of stool (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Blood in urine (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No